CLINICAL TRIAL: NCT03636659
Title: Multi-Center, Open-Label, Randomized, Two Treatment, Parallel, Single Period, Multiple-Dose, Steady State, Global Bioequivalence Study of Amphotericin B Liposome for Injection 50mg /Vial in Patients With Visceral Leishmaniasis
Brief Title: Steady State Global Bioequivalence Study of Amphotericin B Liposome for Injection 50 mg/ Vial in Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aurobindo Pharma Ltd (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR179-17; CTRI/2018/04/013350 (Other: India Council of Medical Research)
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2018-08

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Amphotericin B; liposomal amphotericin B; Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amphotericin B Liposome (Experimental): Amphotericin B Liposome for Injection 50 mg/vial, intravenous infusion at a dose of 3 mg/kg/day, OD for 5 days
  Interventions: Drug: Amphotericin B Liposome
- AmBisome Liposome (Active Comparator): AmBisome Liposome for Injection 50 mg/ vial, intravenous infusion at a dose of 3 mg/kg/day, OD for 5 days
  Interventions: Drug: AmBisome (Amphotericin B) Liposome

INTERVENTIONS:
Drug: Amphotericin B Liposome — Manufactured for: Auromedics Pharma LLC, USA
  Arms: Amphotericin B Liposome
Drug: AmBisome (Amphotericin B) Liposome — Marketed by: Astellas Pharma US, Inc. USA
  Other Names: AmBisome
  Arms: AmBisome Liposome

SUMMARY:
The primary objective is to determine clinical bioequivalence of Amphotericin B liposome for injection of Auromedics Pharma LLC, USA and AmBisome (Amphotericin B) liposome for injection of Astellas Pharma US, Inc., in patients with Visceral Leishmaniasis under fed condition

DETAILED DESCRIPTION:
Multi-Center, Open-Label, Randomized, Two treatment, Parallel, Single period, Multiple-Dose, Steady state, Global Bioequivalence study of Amphotericin B Liposome for Injection 50mg /vial of Auromedics Pharma LLC, USA and AmBisome (Amphotericin B) Liposome for Injection 50mg/vial of Astellas Pharma US, inc. in patients with Visceral Leishmaniasis under fed condition.Sufficient number of patients will be enrolled to have 140 evaluable patients. (90 to 100 patients from India and 40 to 50 patients from Bangladesh).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 18 to 65 years (both inclusive)
* Clinical signs and symptoms of Visceral Leishmaniasis (fever of over 2 weeks duration, weight loss and splenomegaly)
* Presence of amastigotes (Leishmania Donovani bodies) at screening detected by rK39 dipstick test.
* Female subjects of childbearing potential must have a negative serum pregnancy test at enrolment and be willing to use a reliable method of birth control, i.e. barrier method, intrauterine device, or tubal ligation.
* Ability to comply with all study requirements.
* Patients with Hb ≥ 6.0 g/dl
* Patients with platelets count ≥ 60,000/mm3
* Patients should be immunocompetent (e.g., white blood cell count ≥ 2500/ mm3)
* Patients and/ or LAR must be give written informed consent
* Patients with clinically acceptable results from all the screening laboratory parameters and investigations.

Exclusion Criteria:

* Known allergy or hypersensitivity reactions to any components of conventional or liposomal Amphotericin B formulations.
* Any condition which the investigator thinks may prevent the patient from completing the study therapy and subsequent follow-up.
* Pregnant or lactating women
* Patients requiring dose adjustment during the study.
* Serum creatinine concentration greater than twice the upper limit of normal (ULN), AST or ALT value greater than 10 times the ULN
* Patients who are required to be on concomitant therapy with IV fat emulsions, such as total parental nutrition (TPN).
* Patients with total bilirubin levels > 3 times the upper normal limits (i.e. > 3.0 mg/dl).
* Patient with clinically significant Hematopoietic, renal, hepatic and electrolyte disorders (Low level of Magnesium and potassium) will be excluded as per the discretion of Investigator
* Patients with Clinically significant screening laboratory parameters in the opinion of the investigator.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* History of uncontrolled diseases, such as thyroidal dysfunction, angina pectoralis, serious cardiac arrhythmias, serious heart failure, neuropsychiatric infection or disease.
* Patients with controlled and uncontrolled diabetes mellitus
* Patients with Uncontrolled hypertension will be excluded.
* Immunocompromised patients will be excluded from participating the study
* Patients with known positivity for human immunodeficiency virus (HIV), HBsAg and HCV.
* Positive results for drugs of abuse (benzodiazepines, opioids, amphetamines, cannabinoids, cocaine and barbiturates) in urine.
* Positive results for alcohol as detected by alcohol breath analyzer.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* An unusual or abnormal diet, for whatever reason e.g. religious fasting.
* History of donation of blood (1 unit or 350 ml) within 90 days prior to receiving the first dose of investigational medicinal product in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Estimation of Cmax-ss, Maximum concentration over the steady state dosing interval | 05 days
  To establish bioequivalence limits within 80-125 %
Estimation of AUC0-tau, Area under the plasma concentration time curve over the steady state dosing interval | 05 days
  To establish bioequivalence limits within 80-125 %

SECONDARY OUTCOMES:
Evaluation of Cmin-ss | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated
Evaluation of Cavg-ss | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated
Evaluation of tmax-ss | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated
Evaluation of Cpd | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated
Evaluation of Percentage Fluctuation | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated
Evaluation of Swing | 05 days
  Summary statistics, ANOVA, Ratio Analysis, 90% Confidence Interval, Inter subject variability and Power will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nagesh Meda, M.Pharm, Study Chair — Aurobindo Pharma Ltd; Dr. Subhra Lahiri, Ph.D, Study Director — Axis Clinicals Limited; Dr. Sajid Mohd, MD, Study Director — Axis Clinicals Limited; Dr. Krishna Pandey, MD, Principal Investigator — Rajendra Memorial Research Institute of Medical Sciences; Dr. Shyam Sundar, MD, Principal Investigator — Kala-Azar medical Research Centre; Dr. Dinesh Mondal, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research b
Locations (3):
- International Centre for Diarrhoeal Disease Research b, Dhaka, Bangladesh
- India (2):
  - Kala-Azar medical Research Centre, Muzaffarpur, Bihar
  - Rajendra Memorial Research Institute of Medical Sciences, Patna, Bihar

IPD SHARING:
Plan to Share IPD: No